CLINICAL TRIAL: NCT07023874
Title: Dexmedetomidine Combined With Bupivacaine in Ultrasound-guided Pecto-Intercostal Fascial Block in Cardiac Surgery: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Combined With Bupivacaine in Ultrasound-guided Pecto-Intercostal Fascial Block in Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Elbardan, LECTURER OF ANESTHESIA AND SURGICALMINTENSIVE CARE, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0108877
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain; Cardiac Surgery
Keywords: pectointercostal fascial plain block; dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine only in pectointercostal fascial plain block (Active Comparator): Participants will receive bilateral ultrasound-guided pecto-intercostal fascial plane block using 30 mL of 0.25% bupivacaine on each side
  Interventions: Procedure: Bupivacaine group
- bupivacaine and dexmedetomidine in pectointercostal fascial plain block (Experimental): Participants will receive bilateral ultrasound-guided pecto intercostal fascial plane block using 30 mL of 0.25% bupivacaine with one µg/kg dexmedetomidine on each side.
  Interventions: Procedure: bupivacaine + dexmedetomidine group

INTERVENTIONS:
Procedure: Bupivacaine group — Participants will receive bilateral ultrasound-guided pecto-intercostal fascial plane block
  Arms: bupivacaine only in pectointercostal fascial plain block
Procedure: bupivacaine + dexmedetomidine group — Participants will receive bilateral ultrasound-guided pecto intercostal fascial plane block using 30 mL of 0.25% bupivacaine with one µg/kg dexmedetomidine in each side
  Arms: bupivacaine and dexmedetomidine in pectointercostal fascial plain block

SUMMARY:
Recent advancements in pain management techniques suggest that ultrasound-guided peripheral nerve blocks may significantly benefit patients undergoing cardiac surgery. One noteworthy approach is the interfascial thoracic wall plane block, which has become an essential element of multimodal analgesia for post-cardiac surgery care. The pecto-intercostal fascial plane block (PIFPB) is a technique that utilizes ultrasound guidance to administer local anesthetic (LA) into the space between the intercostal muscles and the pectoralis major muscle. This intervention targets the anterior cutaneous branches of the thoracic nerves, particularly T2-T6, which are responsible for sensation in the anteromedial chest wall, including the sternum. Interestingly, the potential role of dexmedetomidine in improving the quality and prolonging the duration of analgesia for post-sternotomy pain through the pecto-intercostal fascial plane block remains unexamined in the current literature, indicating an area ripe for further research.

DETAILED DESCRIPTION:
Optimal management of median sternotomy pain is a critical factor for achieving adequate recovery after cardiac surgery. The mechanisms of postoperative pain related to cardiac surgeries are intricate and multifaceted. The origins of cardiac surgery pain can be neurogenic, musculoskeletal, or visceral. The skin incision, subcutaneous tissue dissection, sternal retraction, preparation of the internal mammary artery graft, placement of chest drains, and sternal wires directly cause tissue injury. Inadequate pain control can potentially be associated with severe adverse effects such as respiratory compromise, increased myocardial work and oxygen demand, delayed mobilisation, and prolonged hospital stay. Further, increased postoperative pain scores are associated with an increased incidence of chronic pain syndromes.

Patient-controlled analgesia with intravenous opioids is most used to alleviate pain after cardiac surgery. Still, opioids can cause adverse effects, including delayed tracheal extubation, respiratory depression, sedation, ileus, nausea, vomiting, immunosuppression, cough suppression, drowsiness and increased risk of chronic pain. Epidural anaesthesia and paravertebral blocks can provide adequate analgesia with earlier extubation and reduced opioid use in cardiac surgical patients. Still, adverse effects related to pneumothorax, injury to the spinal cord, sympathectomy-induced hypotension, and devastating epidural hematoma after full heparinisation have limited their application in cardiac surgical patients.

An ultrasound-guided peripheral nerve block technique may benefit cardiac surgery patients. Interfascial thoracic wall plane blocks have emerged as a valuable component of multimodal analgesia after cardiac surgery. The pecto-intercostal fascial plane block (PIFPB) is an ultrasound-guided parasternal technique that involves the injection of local anaesthetic (LA) into the plane between the intercostal muscles and the pectoralis major muscle. This technique aims to block the anterior cutaneous branches of the thoracic nerves, specifically T2-T6, which innervate the anteromedial chest wall, including the sternum.

A single dose of a local anaesthetic in a peripheral nerve block could provide short-term analgesia, with bupivacaine typically lasting between 4 and 12 hours. Previous studies reported a mean duration of postoperative analgesia after PIFPB ranged from 8 to 12 hours.

Dexmedetomidine had been successfully used with local anaesthetic in peripheral nerve blocks to prolong the duration of analgesia. Dexmedetomidine is a highly selective alpha-2 adrenergic receptor agonist. As an adjuvant to LAs, dexmedetomidine has been the subject of increasing interest because it has the potential to prolong blockade duration. Dexmedetomidine facilitates nerve block through several mechanisms. It inhibits neurons' sodium channels and potassium currents while blocking the hyperpolarization-activated cyclic nucleotide-gated channel, enhancing activity-dependent hyperpolarisation.

The application of dexmedetomidine in enhancing the quality and duration of analgesia for post-sternotomy pain via the pecto-intercostal fascial plane block has yet to be explored in the existing literature. In this study, we hypothesise that dexmedetomidine in conjunction with bupivacaine within an ultrasound-guided PIFPB block may prolong the duration of postoperative analgesia, reduce opioid consumption and achieve better analgesia after sternotomy compared to bupivacaine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Both sexes.
3. ASA physical status class II or III.
4. Elective fast-tracking on-pump cardiac surgery.

Exclusion Criteria:

1. The patient refused to participate in the study.
2. Cognitive impairment or mental disorders.
3. Hepatic and renal impairment.
4. Congestive heart failure.
5. Urgent/emergent surgery.
6. BMI <18 and >35 (kg/m2).
7. Documented allergy to local anaesthetics or dexmedetomidine.
8. Use of chronic pain medications.
9. Previous sternotomy or chest surgery.
10. Patients with a history of substance abuse.
11. Requires the use of mechanical circulatory support pre-operatively.
12. Patients who will not be candidates for fast-tracking extubation after block administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
amount of opioid consumption at 24 hours after ICU admission | 24 hours after ICU admission
  Postoperative total fentanyl consumption: total dose of fentanyl (µg/kg) administered postoperatively during the first postoperative 24 h after ICU admission.

SECONDARY OUTCOMES:
time to extubation | 6 hours after ICU admiision
  Time to extubation (minutes): duration between ICU admission and tracheal extubation
the intensity of postoperative pain at rest and upon coughing | 24 hours after extubation
  The Numeric Rating Scale (NRS) (0-10) will be assessed at rest and cough, with 0 as "no pain," 1-3 as "mild pain," 4-6 as "moderate pain," and 7 10 as "severe pain." If the NRS for pain is more or equal to 4 at any point, then rescue analgesia will be administered. It will be measured immediately after extubation, 2, 4, 8, 12, and 24 hours after extubation.
time to first rescue analgesia | 24 hour after ICU admission
  The time until the first request of fentanyl analgesia is recorded from the ICU admission time.
patient satisfaction | 24 hour after ICU admission
  patient satisfaction with postoperative pain control will be assessed on a four-point scale: Excellent, Good, Fair, and Poor.

CONTACTS AND LOCATIONS:
Overall Officials: LECTURER OF ANESTHESIA AND SURGICAL INTENSIVE CARE, Principal Investigator — University of Alexandria

IPD SHARING:
Plan to Share IPD: No